CLINICAL TRIAL: NCT06405568
Title: Support for Physical Activity for Adults Registered in the Ontario Breast Screening Program: A Randomized Controlled Trial
Brief Title: Physical Activity for Adults in the Ontario Breast Screening Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Cancer Society (CCS) (Other)
Responsible Party: Principal Investigator, Jennifer Brunet, Full Professor, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 156827
Record Dates: First submitted 2024-04-12; First posted 2024-05-08 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer Female; Physical Inactivity
Keywords: Healthcare providers; Physical activity; Breast cancer
MeSH Terms: conditions — Sedentary Behavior; Motor Activity; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The proposed study is a parallel-arm randomized controlled trial. Individuals enrolled in the Ontario Breast Screening Program for High-Risk Screening will be invited by mail to contact research staff who will obtain informed consent. Individuals who self-report engaging in >150 minutes of moderate-to-vigorous intensity physical activity (PA) each week or a condition that makes it unsuitable for participation in this study (e.g., hypertension) will be excluded. Participants will receive a copy of PA recommendations plus a PA motivation package (intervention arm), or just a copy of PA recommendations (control arm); the control arm will receive the PA motivation package after study completion. All participants will complete primary (PA) and secondary (quality of life, BMI) outcome measures at baseline (pre-randomization) and after six weeks online. All outcomes will be analyzed according to intention-to-treat principles according to their randomized allocation and performed using SPSS.
Who Masked: Participant, Investigator
Masking Description: The randomization will be concealed to the investigators throughout the trial; the investigators will not take part in the assessments or intervention delivery. The randomization will be concealed to study staff and participants until informed consent and baseline data are obtained. Study staff will be unblinded to group allocation upon randomization to enable delivery of the intervention arm and control arm corresponding materials, whereas the randomization will remain concealed to participants. To support blinding, all participants will be informed they are being enrolled in a study investigating ways to promote PA and will be kept blind to the fact that the intervention arm receives more materials than the control arm, and thus all (including participants allocated to the control arm) will receive materials (i.e., a copy of PA recommendations). Moreover, we do not anticipate participants to have contact with participants of the other arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical activity recommendations plus motivation package (Intervention Arm) (Experimental): Participants randomized to the intervention arm will receive a package consisting of two components: (1) a copy of age-appropriate physical activity (PA) recommendations matching the Canadian Society of Exercise Physiology (CSEP) recommendations and spotlighting PA benefits, and (2) a PA motivation package including: (a) a link to a website to view three 20-minute webinars covering PA benefits (for cancer risk reduction, quality of life, and weight management) and how to get started using the digitized PA materials and logbook, (b) digitized PA materials containing information explaining and supporting PA recommendations, examples of easy and safe PA participation for all, and activity sheets on behaviour change tools for sustaining PA, and (c) a PA logbook with instructions on how to track PA and tips for increasing PA.
  Interventions: Behavioral: Physical activity intervention
- Standard care and physical activity recommendations (Control Arm) (No Intervention): Participants randomized to the control arm will receive standard care (medical consultations/monitoring at the discretion of each patient's care team) and be advised to continue regular daily living activities; physical activity (PA) restrictions will not be imposed. To facilitate trial retention and because contamination could occur as control arm participants' care team may recommend PA as part of their practice, participants will receive a copy of age-appropriate PA recommendations matching the Canadian Society of Exercise Physiology (CSEP) recommendations and spotlighting PA benefits. This further helps to mitigate the risk that knowledge of which arm a participant has been allocated to leads to moral demoralization in control arm participants. The control arm participants will receive the PA motivation package post-study completion to encourage study completion.

INTERVENTIONS:
Behavioral: Physical activity intervention — Participants will receive a copy of physical activity (PA) recommendations plus a PA motivation package - namely three 20-minute online webinars (explaining PA benefits and how to get started), digitized PA materials (integrating evidence-based behaviour change tools, and a digitized logbook (to track PA).
  Arms: Physical activity recommendations plus motivation package (Intervention Arm)

SUMMARY:
There is "strong" evidence that physical activity (PA) can reduce the risk of breast cancer, which is important for individuals at higher-than-average risk due to their family history or genetic susceptibility. PA can also enhance quality of life (QoL), fitness, and surrogate markers linked to cancer prognosis (e.g., weight). Despite this evidence, most individuals in this cohort are insufficiently active, meaning they do not meet Canadian recommendations of at least 150 minutes of PA each week. This study aims to develop materials that can help increase the number of adults at higher-than-average risk who meet PA recommendations, alongside improving QoL and body mass index (BMI; a measure of one's body weight-height ratio). Participants will include individuals assigned female at birth, aged 30-69 years, at high-risk of breast cancer registered in the Ontario Breast Screening Program who will be randomly assigned to receive (1) the intervention, which includes a copy of PA recommendations (Canadian Society for Exercise Physiology [CSEP] recommendations for adults plus content spotlighting PA benefits) plus a PA motivation package featuring three 20-minute online webinars (explaining PA benefits and how to get started), digitized PA materials (providing evidence-based tools to modify behaviour), and a digitized logbook (to track PA) or (2) only a copy of PA recommendations.

DETAILED DESCRIPTION:
Considerable research (>500 studies) has examined the association between physical (in)activity and cancer incidence. Reviews of observational studies have led to the conclusion that there is some evidence for a reduced risk of 11 different cancer sites when comparing the highest to the lowest levels of physical activity (PA). Specifically, there is "strong" evidence that PA reduces the risk of bladder, breast, colon, endometrial, esophageal adenocarcinoma, and gastric cancers. As a result, public health agencies (e.g., Public Health Agency of Canada) promote PA as an important part of a healthy lifestyle and note that regular PA can help to reduce the risk of premature death and chronic diseases including breast cancer. The Canadian Society for Exercise Physiology (CSEP; https://csepguidelines.ca/guidelines/adults-18-64/) published recommendations for adults (aged 18-64) that include: (a) performing at least 150 minutes of moderate-to-vigorous intensity PA each week (i.e., activities that get your heart beating faster), (b) performing muscle strengthening activities at least twice a week, (c) limiting time spent sitting or laying down to 8 hours or less a day, and (d) achieving good quality and consistent sleep (i.e., 7 to 9 hours, with consistent bed and wake-up times).

Efforts to promote PA in adults at higher-than-average risk for breast cancer (reflected by their enrollment in the Ontario Breast Screening Program), are critical to reduce their risk of breast cancer. Despite the effectiveness of PA recommendations delivered through health care providers (HCPs), most individuals do not receive them during routine care as HCPs report barriers to promoting PA (e.g., inadequate training, lack of time/knowledge). Research needs to focus on developing sustainable interventions that can be implemented broadly using distance-based approaches and available infrastructure (e.g., patient registries) without burdening HCPs to increase the consistency with which PA is promoted to adults at higher-than-average risk for breast cancer. Unlike self-guided PA interventions, supervised face-to-face PA interventions can be costly, unsustainable, and have limited ability to reach individuals unable (or unwilling) to travel to a facility where interventions are delivered. Thus, online interventions should be explored as a means to expand support to adults at higher-than-average risk for breast cancer, as a complement to offering PA recommendations. When self-guided, these interventions are easily scalable at a relatively low marginal cost per additional participant. When self-guided, these interventions are easily scalable at a relatively low marginal cost per additional participant, accessible, self-paced, and available around the clock. Accordingly, they are frequently valued for their accessibility and convenience. Additionally, as interventions incorporating behaviour change techniques, such as goal setting and problem-solving, show greater sustained PA levels post-intervention, it is critical to embed those evidence-based techniques and PA materials (e.g., printed materials, logbook, webinars and education sessions) into online interventions if they are to be effective.

Accordingly, this team of researchers and HCPs have partnered to develop and evaluate an intervention comprising of a copy of PA recommendations for adults (18-64 years) plus a motivation package (intervention arm) that can be implemented using a distance-based approach and sustained in the current healthcare system without burdening HCPs. This study aims to test the following hypothesis: the effects of the intervention on PA (primary outcome), quality of life (QoL) (secondary outcome), and body mass index (BMI; secondary outcome) in adults at high-risk of breast cancer will be greater in comparison to standard care plus a copy of PA recommendations for adults (control arm).

ELIGIBILITY:
Inclusion Criteria:

* English- and French-speaking adults enrolled in the Ontario Breast Screening Program;
* Aged 30-69 years;
* Assigned female at birth;
* Be at high risk for breast cancer as identified through Category A or B, after genetic assessment: (a) Category A individuals meet ≥1 of the following criteria: (i) known carrier of a gene mutation (e.g., BRCA1, BRCA2), (ii) first degree relative of a carrier of a gene mutation (e.g., BRCA1, BRCA2), received genetic counselling but declined genetic testing, (iii) previously assessed as having ≥25% lifetime risk of breast cancer on basis of family history, or (iv) received chest radiation before age 30 and ≥ 8 years previously.

  (b) Category B individuals meet ≥1 of the following criteria: (i) first degree relative of a carrier of a gene mutation (e.g., BRCA1, BRCA2), has not had genetic counselling or testing, (ii) a personal or family history of ≥1 of the following: ≥2 cases of breast cancer and/or ovarian cancer in closely related blood relatives, bilateral breast cancer, both breast cancer and ovarian cancer in the same individual, breast cancer at age ≤35 years, invasive serous ovarian cancer, breast cancer and/or ovarian cancer in Ashkenazi Jewish families, an identified gene mutation (e.g., BRCA1, BRCA2) in any blood relative, male breast cancer.

Exclusion Criteria:

Individuals self-reporting

* >150 minutes of moderate-to-vigorous intensity physical activity in the past week;
* no access to an internet connected device;
* a condition preventing physical activity (e.g., uncontrolled hypertension)

Ages: 30 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Physical activity (PA; aerobic) | Week 0 (baseline) survey and Week 6 survey
  PA will be measured using the Leisure Time Exercise Questionnaire. The questionnaire includes questions on the frequency of light, moderate, and strenuous activities lasting more than 15 minutes during a typical seven-day period. Responses will be aggregated to arrive at one reported value reflecting PA.
Physical activity (PA; strength) | Week 0 (baseline) survey and Week 6 survey
  Participants will be asked to report on their strength and resistance training using a questionnaire created by Principal Investigator Dr. Brunet.

SECONDARY OUTCOMES:
Quality of life (QoL) | Week 0 (baseline) survey and Week 6 survey
  General QoL and specific domains of QoL (i.e., general health perceptions, physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal/emotional problems, emotional well-being, social functioning, energy/fatigue) will be assessed using the RAND 36-Item Short Form Health Survey.
Body Mass Index (BMI) | Week 0 (baseline) survey and Week 6 survey
  Self-report BMI will be computed using two self-reported values (i.e., body mass in kilograms and height in meters) with the following formula: kg/m^2.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Brunet, PhD, Principal Investigator — University of Ottawa

IPD SHARING:
Plan to Share IPD: No
Participants' data will be anonymized using a study identification number (i.e., Participant ID number) that will be stored using a protected file separated from the research data. This file will be stored on a secured Microsoft OneDrive server at the University of Ottawa where only the Provincial Applicant, Dr. Brunet, and study staff/volunteers supervised by Dr. Brunet will have access to the file/research data.

REFERENCES:
- [Background] Friedenreich CM, Ryder-Burbidge C, McNeil J. Physical activity, obesity and sedentary behavior in cancer etiology: epidemiologic evidence and biologic mechanisms. Mol Oncol. 2021 Mar;15(3):790-800. doi: 10.1002/1878-0261.12772. Epub 2020 Aug 18. PMID 32741068
- [Background] McTiernan A, Friedenreich CM, Katzmarzyk PT, Powell KE, Macko R, Buchner D, Pescatello LS, Bloodgood B, Tennant B, Vaux-Bjerke A, George SM, Troiano RP, Piercy KL; 2018 PHYSICAL ACTIVITY GUIDELINES ADVISORY COMMITTEE*. Physical Activity in Cancer Prevention and Survival: A Systematic Review. Med Sci Sports Exerc. 2019 Jun;51(6):1252-1261. doi: 10.1249/MSS.0000000000001937. PMID 31095082
- [Background] McTiernan A, Schwartz RS, Potter J, Bowen D. Exercise clinical trials in cancer prevention research: a call to action. Cancer Epidemiol Biomarkers Prev. 1999 Mar;8(3):201-7. PMID 10090297
- [Background] Patel AV, Friedenreich CM, Moore SC, Hayes SC, Silver JK, Campbell KL, Winters-Stone K, Gerber LH, George SM, Fulton JE, Denlinger C, Morris GS, Hue T, Schmitz KH, Matthews CE. American College of Sports Medicine Roundtable Report on Physical Activity, Sedentary Behavior, and Cancer Prevention and Control. Med Sci Sports Exerc. 2019 Nov;51(11):2391-2402. doi: 10.1249/MSS.0000000000002117. PMID 31626056
- [Background] Hebert ET, Caughy MO, Shuval K. Primary care providers' perceptions of physical activity counselling in a clinical setting: a systematic review. Br J Sports Med. 2012 Jul;46(9):625-31. doi: 10.1136/bjsports-2011-090734. PMID 22711796
- [Background] Haines TP, Sinnamon P, Wetzig NG, Lehman M, Walpole E, Pratt T, Smith A. Multimodal exercise improves quality of life of women being treated for breast cancer, but at what cost? Randomized trial with economic evaluation. Breast Cancer Res Treat. 2010 Nov;124(1):163-75. doi: 10.1007/s10549-010-1126-2. Epub 2010 Aug 24. PMID 20734132
- [Background] Ormel HL, van der Schoot GGF, Sluiter WJ, Jalving M, Gietema JA, Walenkamp AME. Predictors of adherence to exercise interventions during and after cancer treatment: A systematic review. Psychooncology. 2018 Mar;27(3):713-724. doi: 10.1002/pon.4612. Epub 2018 Jan 26. PMID 29247584
- [Background] Sevick MA, Dunn AL, Morrow MS, Marcus BH, Chen GJ, Blair SN. Cost-effectiveness of lifestyle and structured exercise interventions in sedentary adults: results of project ACTIVE. Am J Prev Med. 2000 Jul;19(1):1-8. doi: 10.1016/s0749-3797(00)00154-9. PMID 10865157
- [Background] Brunet J, Wurz A, Nader PA, Belanger M. A systematic review summarizing the effect of health care provider-delivered physical activity interventions on physical activity behaviour in cancer survivors. Patient Educ Couns. 2020 Jul;103(7):1287-1301. doi: 10.1016/j.pec.2020.02.002. Epub 2020 Feb 8. PMID 32067858
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- See also: Physical Activity and Health Promotion Laboratory Official Website — http://www.pahealthpromolab.com